CLINICAL TRIAL: NCT06244459
Title: Virtual Reality Mediated Functional Status Assessment in Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Ahmet Kivanc Menekseoglu, Principal Investigator, Istanbul University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KAEK/2022.11.222
Record Dates: First submitted 2024-01-20; First posted 2024-02-06 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: Hemiplegia
Keywords: virtual reality; assessment
MeSH Terms: conditions — Hemiplegia

STUDY DESIGN:
Intervention Model Description: Participants diagnosed with stroke will be evaluated with the Box and Block Test, 360 degree rotation test and 5 times squat test. These tests will be presented to the participants first in the real world and then in virtual reality.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hemiplegia Group (Experimental): Participants diagnosed with stroke will be evaluated with the Box and Block Test, 360 degree rotation test and 5 times squat test. These tests will be presented to the participants first in the real world and then in virtual reality.
  Interventions: Other: VR Assessment Tool

INTERVENTIONS:
Other: VR Assessment Tool — Participants diagnosed with stroke will be evaluated with the Box and Block Test, 360 degree rotation test and 5 times squat test. These tests will be presented to the participants first in the real world and then in virtual reality.

SUMMARY:
The aim of the study is to investigate the applicability of virtual reality-mediated functional status assessment of patients diagnosed with stroke. Remote assessment of patients and remote rehabilitation (tele-rehabilitation) has an increasing application area in individuals with chronic neurological diseases. In this study, it was aimed to evaluate the upper extremity and balance functions of stroke patients with the developed software.

DETAILED DESCRIPTION:
This prospective and descriptive study will be conducted with patients diagnosed with stroke. Patients diagnosed with stroke will first be evaluated by an expert physiatrist in a clinical setting to determine their functional status, and then evaluated by a virtual reality mediated software system. The evaluation of a patient will take approximately 1 hour.

Participants diagnosed with stroke will be evaluated in terms of hand and balance functions. The measurement parameters planned to be performed are scales routinely applied in stroke patients. Hand functions of the users will be evaluated with the 'Wooden Box and Block Test' , lower extremity muscle strength and fall risk will be evaluated with the 'Sit and Stand Test for 5 Times', and balance functions will be evaluated with the '360 Degree Rotation Test' . The tests mentioned above will be presented to the users first in the real world and then in the virtual reality environment and an objective functional status assessment will be made.

A total of 30 patients diagnosed with stroke are planned to be included in the study.

ELIGIBILITY:
Inclusion Criteria:

* To be between the ages of 18-65,
* History of stroke
* Accept to participate in the study,

Exclusion Criteria:

* Presence of known central nervous system or peripheral nervous system disease other than stroke, presence of progressive neurological deficit,
* Uncontrolled hypertension, diabetes, cardiovascular disease etc.
* Cognitive impairment causing difficulty in performing simple commands
* Epilepsy
* Pregnancy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
Box and Block Test | 1 day
  The Box and Block Test measures unilateral gross manual dexterity. It is calculated how many cubes the patient moves between the compartments in 1 minute with both hands separately.
360 degree rotation test | 1 day
  It is a useful and practical test to evaluate the balance functions of patients. It is calculated how many seconds it takes the patient to complete one full round.
5 times Squat Test | 1 day
  It is performed to evaluate the balance and lower extremity functions of the patients, and the number of seconds it takes to squat 5 times is calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmet Menekseoglu, MD, Principal Investigator — Kanuni Sultan Suleyman Research and Training Hospital
Locations (1):
- Ahmet Kıvanç Menekşeoğlu, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The data obtained as a result of the study will be used within the scope of academic study by protecting the personal information of the participants.

REFERENCES:
- [Result] Mathiowetz V, Volland G, Kashman N, Weber K. Adult norms for the Box and Block Test of manual dexterity. Am J Occup Ther. 1985 Jun;39(6):386-91. doi: 10.5014/ajot.39.6.386. PMID 3160243
- [Result] Mong Y, Teo TW, Ng SS. 5-repetition sit-to-stand test in subjects with chronic stroke: reliability and validity. Arch Phys Med Rehabil. 2010 Mar;91(3):407-13. doi: 10.1016/j.apmr.2009.10.030. PMID 20298832
- [Result] Dite W, Temple VA. Development of a clinical measure of turning for older adults. Am J Phys Med Rehabil. 2002 Nov;81(11):857-66; quiz 867-8. doi: 10.1097/00002060-200211000-00010. PMID 12394998